CLINICAL TRIAL: NCT05061212
Title: The Mechanism of Extracellular Vesicles Containing Mitochondrial DNA in ARDS Lung Injury Caused by Extrapulmonary Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Chun Pan, Department of Critical Care Medicine, Zhongda Hospital, School of Medicine, Southeast University, Southeast University, China
Other Study IDs: ARDS-mtDNA EVs
Record Dates: First submitted 2021-09-18; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The acute respiratory distress syndrome (ARDS) remains a common and morbid complication of critical illness. Sepsis contribute to a lot of ARDS cases, but mechanisms by which non-pulmonary insults such as extrapulmonary sepsis propagate lung injury remain unclear. Most eukaryotic cells release small anuclear membrane-bound vesicles into the extracellular environment in either physiological or pathophysiological conditions, often called extracellular vesicles (EVs) .Through their cargo containing bioactive molecules such as proteins, mRNAs, and microRNAs and their interaction with target cells, EVs are recognized as important mediators of cellular communication. Mitochondrial contents are clearly present in EVs, and mitochondrial cargo within EVs have been shown to stimulate the production of proinﬂammatory cytokines, further enhancing LPS-induced inﬂammation. Among the mitochondrial contents, mtDNA was present at higher levels in EVs.Therefore, we hypothesis, EVs containing mtDNA play an important role in the occurrence and development of ARDS caused by extrapulmonary sepsis.

DETAILED DESCRIPTION:
Inclusion criteria: Patients with ARDS caused by abdominal infection Exclusion criteria: age <18 years old or pregnancy; death or discharge within 24 hours after admission; advanced tumor The pathological information of the patients was collected on 24h, 48h after admission including demographic data, Acute Physiology and Chronic Health Evaluation (APACHE) II score , number of organ failures included in the Sequential Organ Failure Assessment (SOFA) score. The levels of lactate and inflammatory mediators (i.e., plasma C-reactive protein and procalcitonin) were detected on 24h and 48h after admission. All patients were followed up for 28 days, and all-cause mortality was recorded. The durations of mechanical ventilation and ICU stay were also recorded. The primary outcome was mortality on Day 28. Secondary outcomes included the ventilator days and ICU length of stay.

Peripheral blood samples (2 mL) were collected on 24h and 48h after admission to the ICU. EVs were isolated from the plasma, and mtDNA concentration of plasma DNA was evaluated by RT-qPCR.

ELIGIBILITY:
Inclusion Criteria:

Patients with ARDS caused by abdominal infection

Exclusion Criteria:

age <18 years old or pregnancy; death or discharge within 24 hours after admission; advanced tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We enrolled patients with ARDS caused by abdominal infection
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | All patients were followed up for 28 days

SECONDARY OUTCOMES:
Ventilator days | All patients were followed up for 28 days
ICU stay | All patients were followed up for 28 days